CLINICAL TRIAL: NCT00184405
Title: Preventive Peer Groups for Children of Parents With Psychiatric and Addictive Problems (COPP). Child Experiences and Observed Child Changes Following the Intervention
Brief Title: Child Results Following Preventive Children of Parents With Psychiatric and Addictive Problems (COPP) Groups
Status: Terminated | Type: Observational
Why Stopped: Terminated due to financial cut
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Helse Nord-Trøndelag HF (Other)
Responsible Party: Sponsor
Other Study IDs: 4.2005.393
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Psychiatric Disorder NOS
Keywords: Parents with psychiatric or addictive problems
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a study evaluating changes in quality of life and global functioning across and after a manualized peer-group preventive intervention for children of parents with psychiatric or addictive problems.

DETAILED DESCRIPTION:
Self-reported quality of life and based on the group-interviews "ILK" and "Kindl" and general adaptive functioning (CGAS) as reported by teachers and parents will be measured before, after and at follow-up relative to the manualized peer-group preventive intervention. Parents will also complete self-reports on anxiety and depressive symptoms, personality, bonding and attribution before the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Family including Parent with psychiatric or addictive problems

Exclusion Criteria:

* acute severe disorder

Ages: 8 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Families with at least one parent with psychiatric or addictive problem
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2005-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tormod Rimehaug, Asst. Prof., Principal Investigator — Norwegian University of Science and Technology (NTNU), Faculty of Medicine, Dept. of Neuroscience, Center for Child and Adolescent Mental Health
Locations (1):
- Norwegian University of Science and Technology (NTNU), Faculty of Medicine, Dept. of Neuroscience, Center for Child and Adolescent Mental Health, Trondheim, Norway